CLINICAL TRIAL: NCT07165938
Title: Genetics of Neonatal Encephalopathy and Related Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alissa D'Gama, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: IRB-P00051611
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Neonatal Encephalopathy; Hypoxic Ischaemic Encephalopathy (HIE)
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, blood, saliva, buccal, tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonatal Encephalopathy: Individuals with a history of NE who are less than 6 years old at the time of enrollment and available biological parents. Must be followed clinically at Boston Children's Hospital. Research genomic sequencing with CLIA confirmation of diagnostic findings. Those with an existing genetic diagnosis or who are deceased prior to enrollment are ineligible.

SUMMARY:
Investigators at Boston Children's Hospital are conducting research in order to better understand the genetic factors which may contribute to neonatal encephalopathy (NE) and related disorders. These findings may help explain the broad spectrum of clinical features and outcomes seen in individuals with a history of NE.

DETAILED DESCRIPTION:
Neonatal encephalopathy (NE) is a disorder of term newborns involving dysfunction of the central nervous system and can impact one's health throughout the lifespan. While NE can be caused by a number of exposures or external factors, in some cases there is no cause identified or the severity of the condition cannot fully be explained by external factors. In these cases, there is increasing evidence to suggest underlying genetic factors may contribute to NE.

The investigators' research effort is focused on identifying genetic changes (known as "DNA variants") that cause or contribute to NE. By doing so the investigators hope to improve diagnosis and management of NE.

We have two specific aims:

Aim 1: To identify genetic causes of and contributors to NE and related disorders.

Aim 2: To correlate genetic findings with clinical features.

ELIGIBILITY:
Proband Criteria:

Inclusion Criteria:

* Diagnosed with neonatal encephalopathy during the neonatal period as documented in the electronic medical record
* Less than 6 years old at the time of study enrollment
* Patient at Boston Children's Hospital

Exclusion Criteria:

* Genetic cause of NE already identified
* Deceased prior to enrollment

Parent criteria:

Inclusion Criteria:

- Biological parent of eligible proband (see above)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at Boston Children's Hospital and available biological parents
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2035-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 10 years
  The diagnostic yield of genomic sequencing will be calculated as the percentage of enrolled participants with NE who receive a genetic diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical and genomic data may be shared with approved researchers at Boston Children's Hospital and with approved external collaborators.